CLINICAL TRIAL: NCT04085614
Title: Dynamic Coronary Roadmap for Contrast Reduction
Acronym: DCR4Contrast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XCY612-130576
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dynamic Coronary Roadmap group (Experimental): Patients will be treated via standard of care for Percutaneous Coronary Intervention (PCI) with navigation support of Dynamic Coronary Roadmap.
  Interventions: Device: Percutaneous Coronary Intervention (PCI) with Dynamic Coronary Roadmap
- Control group (Active Comparator): Patients will be treated via standard of care for Percutaneous Coronary Intervention (PCI) without navigation support of Dynamic Coronary Roadmap.
  Interventions: Device: Percutaneous Coronary Intervention (PCI) without Dynamic Coronary Roadmap

INTERVENTIONS:
Device: Percutaneous Coronary Intervention (PCI) with Dynamic Coronary Roadmap — Standard of care Percutaneous Coronary Intervention (PCI) with Dynamic Coronary Roadmap
  Arms: Dynamic Coronary Roadmap group
Device: Percutaneous Coronary Intervention (PCI) without Dynamic Coronary Roadmap — Standard of care Percutaneous Coronary Intervention (PCI) without Dynamic Coronary Roadmap
  Arms: Control group

SUMMARY:
The Dynamic Coronary Roadmap is a commercially available product developed by Philips Medical Systems, a Philips Healthcare company. Dynamic Coronary Roadmap is a software medical device intended to provide a real-time and dynamic angiographic roadmap of coronary arteries. The angiographic roadmap is automatically generated from previously acquired coronary angiograms during the same procedure. Dynamic Coronary Roadmap overlays the angiographic roadmap on live 2D fluoroscopic images, thereby assisting the physician in navigating devices, e.g. (guide) wires, catheters, through the coronary arteries.

This is a multi-center, prospective, unblinded, stratified 1:1 randomized controlled trial to assess whether using Dynamic Coronary Roadmap reduces the total iodinated contrast volume related to Percutaneous Coronary Intervention (PCI) compared to the control group without Dynamic Coronary Roadmap.

DETAILED DESCRIPTION:
Primary objective:

• To assess whether using Dynamic Coronary Roadmap reduces the total iodinated contrast volume related to Percutaneous Coronary Intervention (PCI) compared to the control group without Dynamic Coronary Roadmap.

Secondary objective:

• To assess the total number of contrast enhanced cine angiographic X-ray runs (angiograms) related to Percutaneous Coronary Intervention (PCI) in the Dynamic Coronary Roadmap and control group

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing Percutaneous Coronary Intervention (PCI) with a degree of complexity that anticipates the need for more than 25ml of iodinated contrast volume
* Subject has signed informed consent
* Subject is 18 years of age or older, or of legal age to give informed consent per state or national law

Exclusion Criteria:

* Subject undergoing emergency Percutaneous Coronary Intervention (PCI)
* Subject with ST-segment Elevation Myocardial Infarction (STEMI)
* Subject with Chronic Total Occlusion (CTO)
* Subject undergoing PCI for isolated ostial disease of Left Main Coronary Artery (LMCA) or Right Coronary Artery (RCA)
* Subject undergoing Percutaneous Coronary Intervention (PCI) with Optical Coherence Tomography (OCT) support
* Subject undergoing Percutaneous Coronary Intervention (PCI) with rotational or orbital atherectomy
* Subject with Chronic Kidney Disease (CKD) stage V (estimated Glomerular Filtration Rate (eGFR) < 15 ml/min/1.73 m^2)
* Subject with contrast allergy that cannot be adequately pre-medicated
* Subject participates in a potentially confounding drug or device trial during the course of the study.
* Subject is under 18 years of age, or pregnant woman, or breast feeding woman, or meets an exclusion criteria according to national law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Escaned, MD, Principal Investigator — San Carlos Hospital Madrid
Locations (6):
- United States (2):
  - University of Colorado Hospital, Denver, Colorado
  - Columbia University Medical Center/NYPH, New York, New York
- Grand Hôpital de Charleroi Saint-Joseph, Charleroi, Belgium
- Hadassah Medical Center, Jerusalem, Israel
- Spain (2):
  - San Carlos Hospital, Madrid
  - Fuenlabrada University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hennessey B, Danenberg H, De Vroey F, Kirtane AJ, Parikh M, Karmpaliotis D, Messenger JC, Strobel A, Curcio A, van Mourik MS, Eshuis P, Escaned J. Dynamic Coronary Roadmap versus standard angiography for percutaneous coronary intervention: the randomised, multicentre DCR4Contrast trial. EuroIntervention. 2024 Feb 5;20(3):e198-e206. doi: 10.4244/EIJ-D-23-00460. PMID 38343370
- [Derived] Hennessey B, Messenger JC, Kirtane AJ, Parikh M, Danenberg H, De Vroey F, Curcio A, Eshuis P, Escaned J. Rationale and design of the Dynamic Coronary Roadmap for Contrast Reduction (DCR4Contrast) in PCI randomized controlled trial. Am Heart J. 2023 Sep;263:151-158. doi: 10.1016/j.ahj.2023.04.004. Epub 2023 Apr 9. PMID 37040861

RESULTS

PARTICIPANT FLOW:
Groups:
- Dynamic Coronary Roadmap Group: Patients will be treated via standard of care for PCI (Percutaneous Coronary Intervention) with navigation support of Dynamic Coronary Roadmap.
  PCI (Percutaneous Coronary Intervention) with Dynamic Coronary Roadmap: Standard of care PCI (Percutaneous Coronary Intervention) with Dynamic Coronary Roadmap
- Control Group: Patients will be treated via standard of care for PCI (Percutaneous Coronary Intervention) without navigation support of Dynamic Coronary Roadmap.
  PCI (Percutaneous Coronary Intervention) without Dynamic Coronary Roadmap: Standard of care PCI (Percutaneous Coronary Intervention) without Dynamic Coronary Roadmap
Period: Overall Study
Arm/Group | Dynamic Coronary Roadmap Group | Control Group
Started | 188 | 183
Completed | 179 | 177
Not Completed | 9 | 6
Not completed — Protocol Violation | 9 | 6

BASELINE CHARACTERISTICS:
Population: The Full Analysis Population (FAP) was defined as all randomized subjects who underwent a Percutaneous Coronary Intervention (PCI) in at least one vessel without the use of Optical Coherence Tomography (OCT) and/or rotational or orbital atherectomy of which the primary endpoint and/or the secondary endpoint were available.
Groups:
- Dynamic Coronary Roadmap Group: Patients will be treated via standard of care for PCI with navigation support of Dynamic Coronary Roadmap.
  PCI with Dynamic Coronary Roadmap: Standard of care PCI with Dynamic Coronary Roadmap
- Control Group: Patients will be treated via standard of care for PCI without navigation support of Dynamic Coronary Roadmap.
  PCI without Dynamic Coronary Roadmap: Standard of care PCI without Dynamic Coronary Roadmap
- Total: Total of all reporting groups
Arm/Group | Dynamic Coronary Roadmap Group | Control Group | Total
Number analyzed (Participants) | 179 | 177 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (10.8) | 65.9 (10.9) | 65.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 143 | 139 | 282
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Self-reported Race: Black or African American | 3 | 6 | 9
  Self-reported Race: Non-Black/Non-African American | 113 | 107 | 220
  Self-reported Race: Unknown | 63 | 64 | 127
Region of Enrollment [Number; unit: participants]
  Belgium | 47 | 47 | 94
  United States | 63 | 57 | 120
  Israel | 46 | 47 | 93
  Spain | 23 | 26 | 49
Weight (kg) [Mean (Standard Deviation); unit: kg] | 85.1 (20.0) | 83.1 (15.6) | 84.1 (18.0)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (5.7) | 28.5 (4.8) | 28.7 (5.2)
Diabetes Mellitus [Count of Participants; unit: Participants] | 66 | 68 | 134
Hypertension (> 140/90 mmHg) [Count of Participants; unit: Participants] | 135 | 124 | 259
Chronic Kidney Disease [Count of Participants; unit: Participants] | 18 | 26 | 44
Prior revascularization [Count of Participants; unit: Participants] | 62 | 60 | 122
Coronary Artery Bypass Graft [Count of Participants; unit: Participants] | 12 | 15 | 27
Prior Myocardial Infarction [Count of Participants; unit: Participants] | 55 | 54 | 109
Severe Left ventricular ejection fraction (<30%) [Count of Participants; unit: Participants] | 2 | 6 | 8
eGFR, ml/min/1.73m^2 [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 77.5 (19.7) | 75.5 (19.9) | 76.5 (19.8)

OUTCOME MEASURES:

1. Primary Outcome: Total Percutaneous Coronary Intervention (PCI) Iodinated Contrast Volume
Description: Average total undiluted contrast volume (in ml, measured by an automatic contrast injector) per Percutaneous Coronary Intervention (PCI), where the start of the PCI is marked by the moment the interventional guiding catheter is positioned in a stable coronary position and the end of the PCI is marked by time of the last PCI check exposure run (angiogram).
Time Frame: During Percutaneous Coronary Intervention (PCI) procedure
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Dynamic Coronary Roadmap Group | Control Group
Number analyzed (Participants) | 179 | 177
ml | 64.6 (44.4) | 90.8 (55.4)

2. Secondary Outcome: Number of Angiograms
Description: Average total number of contrast enhanced cine angiographic X-ray runs (angiograms) per Percutaneous Coronary Intervention (PCI) (from start of PCI marked by the moment the interventional guiding catheter is positioned in a stable coronary position till the end of the PCI marked by the time of the last PCI check exposure run, i.e., angiogram) determined via visual assessment (e.g., on the Philips X-ray system).
Time Frame: During Percutaneous Coronary Intervention (PCI) procedure
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Number of runs
Arm/Group | Dynamic Coronary Roadmap Group | Control Group
Number analyzed (Participants) | 179 | 177
Number of runs | 8.7 (4.7) | 11.7 (7.6)

ADVERSE EVENTS:
Time Frame: Patients were followed-up until discharge through study completion, which was 1 day on average.
Arm/Group | Dynamic Coronary Roadmap Group | Control Group
All-Cause Mortality (participants affected / at risk) | 1/179 | 0/177
Serious Adverse Events (participants affected / at risk) | 14/179 | 7/177
Other Adverse Events (participants affected / at risk) | 0/179 | 0/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dynamic Coronary Roadmap Group (N=179) | Control Group (N=177)
Acute Myocardial Infarction (Cardiac disorders) | 14 (14) | 7 (7) — All Acute Myocardial Infarctions occurred pre study PCI procedure (i.e. unrelated to study participation).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT04085614/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04085614/SAP_001.pdf